CLINICAL TRIAL: NCT07364734
Title: Epidemiological Characteristics and Efficacy Evaluation of Refractory Crohn's Disease: a Multicenter, Prospective and Observational Cohort Study
Brief Title: Epidemiological Characteristics and Efficacy Evaluation of Difficult-To-Treat Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Xiang Gao (Other)
Responsible Party: Sponsor-Investigator, Xiang Gao, Director of Gastroenterology, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2025-ZSLYEC-556
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
Keywords: Difficult-To-Treat Crohn's Disease; Epidemiological Characteristics; Efficacy Evaluation
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total study population: The total study population included all CD patients who visited the Sixth Affiliated Hospital of Sun Yat sen University during the specified time period (November 2025 to January 2026), including newly diagnosed and previously diagnosed patients

SUMMARY:
Difficult to treat Crohn's disease (DTT-CD) was defined by the International Organization for the Study of Inflammatory Bowel Diseases (IOIBD) in 2023, which refers to CD patients with poor response to drug treatment and poor prognosis. Foreign epidemiological studies have shown that DTT-CD accounts for 24.8% of all CD patients, and most of them are patients with advanced treatment failure according to more than two different mechanisms. Our previous retrospective data suggested that compared with foreign DTT-CD patients, there was no significant difference in the proportion of patients with advanced treatment failure due to more than two different mechanisms, but the proportion of patients with recurrence after two intestinal resection and complex anal fistula was increased. Therefore, this project aims to determine the current prevalence and epidemiological status of DTT-CD in China; To clarify the difference in efficacy and prognosis between DTT-CD patients and non DTT-CD patients using advanced treatment (including biological agents and small molecule drugs); Objective to evaluate the incidence and risk factors of non DTT-CD patients progressing to DTT-CD within 1 year. To further verify whether the domestic DTT-CD population is significantly different from the foreign population, and provide theoretical support for the selection of subsequent treatment options.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Crohn's disease was confirmed;
* Patients aged 18-65;
* Informed consent was obtained voluntarily.

Exclusion Criteria:

* The diagnosis of CD was unclear;
* The clinical baseline data were missing seriously;
* Patients currently enrolled in clinical trials or receiving experimental drugs;
* Other contraindications to biologics or small molecule drugs (including active infection, pregnancy, etc.);
* Patients with short bowel syndrome;
* Patients with a small bowel or colostomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease who visited tertiary hospitals, including those newly diagnosed and those previously diagnosed.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
steroid-free remission | From the beginning of enrollment to 1 year
  Compare the steroid-free clinical remission rates of patients with DTT-CD and non DTT-CD during the induction and maintenance periods in the patients using biologics or small molecule drugs. "Steroid-free" refers to patients who do not receive concomitant steroid medication.

SECONDARY OUTCOMES:
Epidemiological status of Difficult-To-Treat Crohn's Disease | From the beginning of enrollment to three months later
  Calculate the proportion of DTT-CD patients in the total population
Clinical reponse rate | From the begining of enrollment to 1 year.
  Compare the clinical response rates of patients with DTT-CD and non DTT-CD during the induction and maintenance periods in the patients using biologics or small molecule drugs.
Clinical remission rate | From the begining of enrollment to 1 year
  Compare the clinical remission rates of patients with DTT-CD and non DTT-CD during the induction and maintenance periods in the patients using biologics or small molecule drugs.
Endoscopic outcome | From the begining of enrollment to 1 year
  Compare the endoscopic outcomes of patients with DTT-CD and non DTT-CD during the induction and maintenance periods, including the endoscopic response rate, the endoscopic remission rate, and the mucusal healing rate in the patients using biologics or small molecule drugs.
Ultrasound outcome | From the begining of enrollment to 1 year
  Compare the ultrasound outcomes of patients with DTT-CD and non DTT-CD during the induction and maintenance periods in the patients using biologics or small molecule drugs, including the transmural response rate and the transmural remission rate.
Postoperative recurrence rate | From the begining of enrollment to 1 year
  Compare the postoperative recurrence rates of DTT-CD and non DTT-CD: postoperative recurrence is defined as the recurrence of clinical symptoms, or endoscopic mucosal ulcers, or imaging evidence of intestinal inflammation, etc.
Safety differences | From the begining of enrollment to 1 year
  Compare the safety differences between DTT-CD and non-DTT-CD after one year of biologic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided